CLINICAL TRIAL: NCT02975726
Title: Peritoneal Dialysis Catheters for the Treatment of Refractory Ascites Management: A Randomized Un-Blinded Pilot Study
Brief Title: Peritoneal Dialysis Catheters for the Treatment of Refractory Ascites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Paul Komenda, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2014:066
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Liver Cirrhosis; Ascites
Keywords: Liver Cirrhosis; Refractory ascites; PD catheter
MeSH Terms: conditions — Liver Cirrhosis; Ascites | interventions — Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peritoneal Dialysis Catheter Insertion (Experimental): Catheters will be inserted at the bedside in a special procedure room.Argyle PD catheter kits will be used:2 cuffed curled catheters at 57cm or 62cm lengths. At time of PD catheter insertion,most patients will be drained of 5-10L of ascites or more to decrease the chance of catheter leaks.The volume removed will be at sole discretion of physician doing the procedure.Patients will be administered 25% Human Serum Albumin injection: 100cc after the 5-10L drainage,and 200cc if 10-15L is removed.Patients will undergo an initial drain and training with a specialized nurse.Patients in this arm will be instructed to drain a maximum of 2L per day after the initial drain.Monthly bloodwork will be performed.
  Interventions: Device: Peritoneal Dialysis Catheter; Biological: 25% Human Serum Albumin injection; Procedure: Bloodwork
- Large Volume Paracentesis (Active Comparator): Patients in this arm of the study will continue their usual practice of LVP as required. They will continue to undergo their LVP procedures through their regular means.Monthly bloodwork will be performed.
  Interventions: Procedure: Large Volume Paracentesis; Procedure: Bloodwork

INTERVENTIONS:
Device: Peritoneal Dialysis Catheter — Peritoneal dialysis catheter insertion in order to drain access fluid within the belly for patients with liver cirrhosis and refractory ascites.
  Arms: Peritoneal Dialysis Catheter Insertion
Procedure: Large Volume Paracentesis — Insertion of a needle into the peritoneal cavity where ascites accumulates, then attaching the needle to a collection system that drains the ascites by gravity. This procedure is part of the standard care for the treatment of refractory ascites.
  Arms: Large Volume Paracentesis
Biological: 25% Human Serum Albumin injection — Patients will be given Human Serum Albumin after the initial drain of ascites fluid: 100cc for 5-10L drainage, 200cc for 10-15L drainage.
  Arms: Peritoneal Dialysis Catheter Insertion
Procedure: Bloodwork — Monthly bloodwork will be done as part of usual standard of care.

SUMMARY:
One complication of liver disease is the buildup of fluid within the belly. This is known as ascites. Patients who have ascites have a decreased appetite, pain, nausea and shortness of breath. Ascites is typically treated with medications, however when that does not work, patients need a procedure where a needle is inserted in the belly every few weeks to drain the excess fluid. About 2 in 5 patients with ascites from liver failure can get kidney disease from their worsening liver function or from the drainage of fluid with needles. Once patients have both advanced liver disease and kidney disease, their chance of dying largely increases.

The present study will be the first of its kind to study a new technique to treat ascites. Investigators are planning to place a tube in a patient's belly to drain the excessive amounts of fluid. This technique is similar to how one type of dialysis is done to treat patients with kidney failure. This study is set as a pilot investigation in order to determine the feasibility of doing a larger, randomized clinical trial investigating the use of this novel technique. Importantly, advanced liver disease patients are at high risk to develop kidney disease, and therefore are an important group to focus on. Investigators believe that this technique will prevent or slow the development of kidney disease in liver failure patients, and improve their quality of life, far more than the current available treatments.

DETAILED DESCRIPTION:
Refractory ascites is when fluid recurrently accumulates in the peritoneal cavity, as an end result of multiple mechanisms, including liver cirrhosis, peritoneal infiltration by tumor, portal hypertension, lymphangitic carcinomatosis, congestive heart failure, or lymphatic obstruction. It is associated with increased mortality and morbidity, including complications of abdominal wall hernias, spontaneous bacterial peritonitis, kidney dysfunction, and pleural effusions. The development of ascites also leads to multiple symptoms including anorexia, early satiety, nausea and vomiting, shortness of breath, and limited mobility.

The management of ascites associated with liver dysfunction usually follows a stepwise escalation in treatments. The initial management typically involves sodium restriction and diuretic therapy up to a daily maximum of 160 mg of furosemide and 400 mg of spironolactone. When ascites no longer can be controlled by these measures, one option is to decrease portal hypertension, a main pathogenic factor in ascites development, by undergoing a procedure called transjugular intrahepatic portosystemic shunt (TIPS). This procedure requires certain patient criteria to be fulfilled and is associated with complications and increased risk of hepatic encephalopathy, and therefore is confined to a small subgroup of patients with ascites. Consequently, abdominal large volume paracentesis (LVP) is the treatment of choice in many patients. This procedure involves insertion of a needle into the peritoneal cavity where ascites accumulates, then attaching the needle to a collection system that drains the ascites by gravity. The definitive treatment for ascites in patients with cirrhosis is a liver transplant, but due to limited supply of organs, and contraindications to transplantation, patients often undergo repeated LVP while waiting on the wait list or until death. Paracentesis is associated with risks including post paracentesis circulatory dysfunction leading to hyponatremia, kidney dysfunction, viscus puncture, and peritonitis. It also is a costly, resource intense, and at times an uncomfortable treatment for patients due to the procedure itself and the need for repeated treatments.

A potential alternative to LVP is the placement of an intraperitoneal catheter, in the same manner that a peritoneal dialysis (PD) catheter, to drain ascites. The procedure has a high technical insertion success rate with minimal complications and is routinely done at the bedside by nephrologist under local anesthesia. PD catheter placement for ascites drainage has many potential advantages, including the ability for it to be done at home by the patient and avoid visits to clinics or hospitals; the frequency of drainage can be timed to patient symptoms, and perhaps have less complication rates than LVP. However, the efficacy and safety of this approach in decompensated cirrhosis when compared to periodic LVP (current standard of care) has not been tested in a randomized trial. Investigators propose a single center, multi-site randomized control trial comparing bedside PD catheter placement versus usual standard of serial LVP for treatment of refractory ascites. The primary outcomes will be improvement of 10 points in the physical component score (PCS) of the Short Form-36 (SF-36) at two months. Investigators plan to randomize 50 patients (25 per arm) based on a power calculation to achieve an 10 point improvement in the PCS-SF-36 (SE = 5). Secondary outcomes will include incidence of mechanical and infectious complications, emergency department utilization, hospitalization and mortality, all other domains of the SF-36, Euroquol-5D (EQ-5D), the Newcastle Patient Reported Ascites Measure and overall health care costs.

Primary Hypothesis: Drainage of ascites associated with liver failure via PD catheter is superior to serial LVP in improving the physical component of quality of life as measured by SF-36.

This trial will be pivotal in possibly changing the standard of care for the management of refractory ascites from cirrhosis. If the primary hypothesis is confirmed, investigators will design and conduct subsequent trials to address potential morbidity and mortality benefits associated with this technique for ascites management.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females greater than 18 years of age.
2. Liver cirrhosis as defined by a histological, clinical, or radiological criteria
3. Patients with refractory non-malignant ascites requiring 2 or more LVPs in the last 4 months.
4. No contraindication for bedside PD catheter insertion (e.g. prior major abdominal surgery, ostomies, large hernias, bleeding diatheses, inability to lie flat).
5. Patients having a support person (family member/friend/caregiver, etc) willing to go through training and help with catheter care.

Exclusion Criteria:

1. Prior liver transplant
2. Is actively being worked up for liver transplant or is already on the liver transplant waitlist
3. Current SBP (spontaneous bacterial peritonitis) defined as polymorphonuclear (PMN) cell count of >250 cells/mm3 in the ascites or positive bacteria in ascitic cultures
4. Malignant ascites
5. Severe coagulopathy with either an INR (international normalized ratio) > 1.5, a platelet count < 50 x 109/L that is not able to be reversed at time of PD catheter insertion
6. Any previous episodes of spontaneous bacterial peritonitis.
7. Loculated ascites
8. Known presence of HIV/AIDS
9. Immunomodulatory treatments used within the last 4 months
10. Expected survival <6 months and/or MELD (The Model for End-Stage Liver Disease) score > 30
11. Hepatic Encephalopathy episode requiring hospital admission in the past 6 months.
12. History of non-compliance or suspected failure to comply with study requirements
13. Allergies to Vancomycin and Cephalosporins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in the physical component of Quality of Life | 2 months post intervention
  Change in the physical component summary score of the SF 36 questionnaire.

SECONDARY OUTCOMES:
Catheter Insertion Technical Success Rate | Day of insertion of PD catheter
  Technical success rate of tunneled PD catheters: Defined as successful positioning of the catheter in the intraperitoneal space with initial drainage of ascites
PD Catheter Survival | Number of days between catheter insertion and possible complication, up to 6 months
  Defined as days from insertion to date of a PD catheter related complication if they occur, assessed during the study timeframe.
PD Catheter Related Complications Frequency | through study completion, up to 6 months
  The number of participants with following complications: 1) Infection at the exit site or tunnel (as defined by the International Society of peritoneal Dialysis 2010 guidelines). 2) Peritonitis 3) intra-luminal/extra-luminal obstruction 4) catheter mal positioning (migration, omental wrapping) 5) Catheter leakage
Large Volume Paracentesis Complications Frequency | through study completion, up to 6 months
  The number of participants with following complications: 1) Peritonitis 2) leakage at puncture site 3) visceral puncture
Participant Self-Reported Health Status | 0,2,4 and 6 months
  Measured by the number of points as a result of participants' answers to SF-36 questionnaire
Participant Health State Description and Evaluation | 0,2,4 and 6 months
  Measured by the number of points as a result of participants' answers to EQ-5D questionnaire
The Impact of Ascites on Health Related Quality of Life | 0,2,4 and 6 months
  Measured by the number of points as a result of participants' answers to Newcastle Patient Reported Ascites Measure questionnaire
Renal Dysfunction Assessment | Monthly, up to 6 months
  Measured by blood work: serum creatinine, serum sodium, potassium, chloride, bicarbonate, urea, glucose, eGFR (estimated glomerular filtration rate).
Renal Function Assessment | at 0 and 6 months
  Measured by 24 hour urine collection: creatinine clearance, urine volume and urine sodium.
Serum Albumin and PD Fluid Albumin Assesment | At 0, 2, and 6 months
  PD catheter arm: Assessment of serum albumin and measurement of albumin in PD fluid at 0, 2, and 6 months
Patient Heart Rate | At regular clinic appointments, through study completion, up to 6 months
  Patient heart rate taken as part of regular physical assessment
Patient Blood Pressure | At regular clinic appointments, through study completion, up to 6 months
  Patient blood pressure taken as part of regular physical assessment
Patient Weight | At regular clinic appointments, through study completion, up to 6 months
  Patient weight taken as part of regular physical assessment
Hospital Visits | through study completion, up to 6 months
  The number of hospital admissions or emergency department visits from complications related to cirrhosis (encephalopathy, gastrointestinal bleed) or peritonitis.
Total Health Care Costs | through study completion, up to 6 months
  Direct health care costs will be estimated for both groups of patients taking a health care payor perspective.
Cost Effectiveness | through study completion, up to 6 months
  A decision analysis, Markov model will be constructed between the two intervention arms with outcomes expressed as cost per quality adjusted live year (cost per QALY) and expressed as incremental cost effectiveness ratios (ICER's).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Komenda, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senousy BE, Draganov PV. Evaluation and management of patients with refractory ascites. World J Gastroenterol. 2009 Jan 7;15(1):67-80. doi: 10.3748/wjg.15.67. PMID 19115470
- [Background] Planas R, Montoliu S, Balleste B, Rivera M, Miquel M, Masnou H, Galeras JA, Gimenez MD, Santos J, Cirera I, Morillas RM, Coll S, Sola R. Natural history of patients hospitalized for management of cirrhotic ascites. Clin Gastroenterol Hepatol. 2006 Nov;4(11):1385-94. doi: 10.1016/j.cgh.2006.08.007. PMID 17081806
- [Background] Singhal S, Baikati KK, Jabbour II, Anand S. Management of refractory ascites. Am J Ther. 2012 Mar;19(2):121-32. doi: 10.1097/MJT.0b013e3181ff7a8b. PMID 21192246
- [Background] Runyon BA; AASLD Practice Guidelines Committee. Management of adult patients with ascites due to cirrhosis: an update. Hepatology. 2009 Jun;49(6):2087-107. doi: 10.1002/hep.22853. No abstract available. PMID 19475696
- [Background] Van Thiel DH, Moore CM, Garcia M, George M, Nadir A. Continuous peritoneal drainage of large-volume ascites. Dig Dis Sci. 2011 Sep;56(9):2723-7. doi: 10.1007/s10620-011-1792-x. Epub 2011 Jul 7. PMID 21735084
- [Background] Peltekian KM, Wong F, Liu PP, Logan AG, Sherman M, Blendis LM. Cardiovascular, renal, and neurohumoral responses to single large-volume paracentesis in patients with cirrhosis and diuretic-resistant ascites. Am J Gastroenterol. 1997 Mar;92(3):394-9. PMID 9068457
- [Background] Lungren MP, Kim CY, Stewart JK, Smith TP, Miller MJ. Tunneled peritoneal drainage catheter placement for refractory ascites: single-center experience in 188 patients. J Vasc Interv Radiol. 2013 Sep;24(9):1303-8. doi: 10.1016/j.jvir.2013.05.042. Epub 2013 Jul 19. PMID 23876552
- [Background] Savin MA, Kirsch MJ, Romano WJ, Wang SK, Arpasi PJ, Mazon CD. Peritoneal ports for treatment of intractable ascites. J Vasc Interv Radiol. 2005 Mar;16(3):363-8. doi: 10.1097/01.RVI.0000147082.05392.2B. PMID 15758132
- [Background] Tapping CR, Ling L, Razack A. PleurX drain use in the management of malignant ascites: safety, complications, long-term patency and factors predictive of success. Br J Radiol. 2012 May;85(1013):623-8. doi: 10.1259/bjr/24538524. Epub 2011 Mar 22. PMID 21427184
- [Background] Barnett TD, Rubins J. Placement of a permanent tunneled peritoneal drainage catheter for palliation of malignant ascites: a simplified percutaneous approach. J Vasc Interv Radiol. 2002 Apr;13(4):379-83. doi: 10.1016/s1051-0443(07)61740-0. PMID 11932368
- [Background] Belfort MA, Stevens PJ, DeHaek K, Soeters R, Krige JE. A new approach to the management of malignant ascites; a permanently implanted abdominal drain. Eur J Surg Oncol. 1990 Feb;16(1):47-53. PMID 1689678
- [Background] Monsky WL, Yoneda KY, MacMillan J, Deutsch LS, Dong P, Hourigan H, Schwartz Y, Magee S, Duffield C, Boak T, Cernilia J. Peritoneal and pleural ports for management of refractory ascites and pleural effusions: assessment of impact on patient quality of life and hospice/home nursing care. J Palliat Med. 2009 Sep;12(9):811-7. doi: 10.1089/jpm.2009.0061. PMID 19622018
- [Background] Fleming ND, Alvarez-Secord A, Von Gruenigen V, Miller MJ, Abernethy AP. Indwelling catheters for the management of refractory malignant ascites: a systematic literature overview and retrospective chart review. J Pain Symptom Manage. 2009 Sep;38(3):341-9. doi: 10.1016/j.jpainsymman.2008.09.008. Epub 2009 Mar 28. PMID 19328648
- [Background] Nessim SJ, Bargman JM, Jassal SV, Oliver MJ, Na Y, Perl J. The impact of transfer from hemodialysis on peritoneal dialysis technique survival. Perit Dial Int. 2015 May-Jun;35(3):297-305. doi: 10.3747/pdi.2013.00147. Epub 2013 Dec 1. PMID 24293665
- [Background] Wong F. Management of ascites in cirrhosis. J Gastroenterol Hepatol. 2012 Jan;27(1):11-20. doi: 10.1111/j.1440-1746.2011.06925.x. PMID 21916992